CLINICAL TRIAL: NCT01100294
Title: Tolerability and Safety Study of FLUVAL P Monovalent Influenza Vaccine in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fluart Innovative Vaccine Ltd, Hungary (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FLUVAL P-H-08
Record Dates: First submitted 2010-03-30; First posted 2010-04-08 (Estimated); Last update posted 2012-05-21 (Estimated); Status verified 2012-05

CONDITIONS: Influenza
Keywords: Influenza; Pandemic vaccine; Seasonal vaccine; Prevention; Influenza vaccine; Influenza in humans; Pandemic influenza in humans; Influenza vaccine for children
MeSH Terms: conditions — Influenza, Human | interventions — Vaccination; Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vaccination with Fluval P (Experimental): Vaccination with Fluval P monovalent influenza vaccine with 6 μg HA/0.5 ml active ingredient content and aluminium phosphate gel adjuvant. Dose: 0.25 ml (total 3 μg HA), single dose.
  Interventions: Biological: Vaccination with FLUVAL P

INTERVENTIONS:
Biological: Vaccination with FLUVAL P — Vaccination with Fluval P monovalent influenza vaccine with 6 μg HA/0.5 ml active ingredient content and aluminium phosphate gel adjuvant.
  Dose: 0.25 ml (total 3 μg HA), single dose.
  Other Names: Influenza; Pandemic vaccine; Prevention; Influenza vaccine; Influenza in humans; Vaccination of children

SUMMARY:
To determine the tolerability and safety of FLUVAL P monovalent influenza vaccine in children.

DETAILED DESCRIPTION:
This is an open, uncontrolled study to assess safety and tolerability of Fluval P monovalent influenza vaccine (whole virus, inactivated, adjuvanted with alumn phosphate gel) containing 6 mcgHA per 0.5mL active ingredient in children of 6-36 months of age. The vaccination is not repeated.

Tolerability and safety (incidence of adverse events) of the study drug is assessed after Day 28 then after Day 180-210 following the vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 to 36 months, both sexes;
* Are in good health (as determined by vital signs and existing medical condition) or are in stable medical condition. Subjects will not be excluded with known adequately treated clinically significant organ or systemic diseases (e.g. asthma or diabetes), such that, in the opinion of the investigator, the significance of the disease will not compromise the subject's participation in the study;
* Capability of the legitimate representative of the volunteer to understand and comply with planned study procedures;
* Legitimate representative of the volunteer provide written informed consent prior to initiation of study procedures;
* Absence of existence of any exclusion criteria.

Exclusion Criteria:

* Known allergy to eggs or other components of the vaccine (in particular mercury);
* History of Guillain-Barré syndrome;
* Active neoplasm;
* Former or on-going immunosuppressive therapy;
* Concomitant corticosteroid therapy, including high-dose inhaled corticosteroids;
* Immunoglobulin (or similar blood product) therapy within 3 months prior to vaccination;
* Documented HIV, HBV or HCV infection;
* Chronic illness that, in the opinion of the investigator, may have effect on the participation in the study;
* Acute febrile respiratory illness within one week prior to vaccination;
* Vaccine therapy within 4 weeks prior to vaccination;
* Influenza vaccination within 6 months prior to vaccination;
* Experimental drug therapy within 1 month prior to vaccination;
* Past or current psychiatric disease of the legitimate representative that upon judgement of the investigator may have effect on the objective decision-making of the legitimate representative;
* Alcohol or drug abuse of the legitimate representative.

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2009-09; Primary Completion 2010-04 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | 28 days after vaccination
  To assess tolerability/safety (incidence of adverse events) of the study drug after Day 28 following the vaccination.

SECONDARY OUTCOMES:
Incidence of adverse events | 180-210 days after vaccination
  To assess safety of the study drug after Day 180-210 following the vaccination.
Efficacy of the study drug | 180-210 days after vaccination
  To assess the efficacy of the study drug by epidemiological follow-up of the participants until Day 180-210 following the vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Ősi, Dr., Study Director — Omninvest Ltd.; Éva Szabó, MD, Principal Investigator — "Csolnoky Ferenc" Veszprém County Hospital
Locations (1):
- "Csolnoky Ferenc" Veszprém County Hospital, Veszprém, Veszprém megye, Hungary